CLINICAL TRIAL: NCT05662254
Title: PERsonalized Mood Augmentation Trial for Depressed Mood
Acronym: PERMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Jyoti Mishra, Associate Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PERMA
Record Dates: First submitted 2022-12-10; First posted 2022-12-22 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Personalized Behavioral Intervention (Experimental): Behavioral lifestyle intervention assigned according to each participant's mood and lifestyle data patterns.
  Interventions: Behavioral: Personalized Behavioral Intervention

INTERVENTIONS:
Behavioral: Personalized Behavioral Intervention — Behavioral lifestyle intervention assigned according to each participant's mood and lifestyle data patterns.

SUMMARY:
The goal of this open-label single-arm study is to test personalized behavioral intervention for depressed mood.

DETAILED DESCRIPTION:
The goal of this open-label single-arm study is to test personalized behavioral intervention for depressed mood. After an initial period (2-4 weeks) of mood and lifestyle monitoring using smartphone and smartwatch data, participants will be assigned to an evidenced-based behavioral plan that target their lifestyle for 6 weeks. The trial will evaluate changes in depressed mood, associated health behaviors and cognition.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate depression per PHQ9 symptom ratings

Exclusion Criteria:

* active substance abuse/dependence
* psychotic disorders
* bipolar disorder
* eating disorder
* displaying acutely suicidal behaviors

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-10-11 (Actual)

PRIMARY OUTCOMES:
PHQ9 | 12 weeks
  Depression Symptoms on the Patient Health Questionnaire 9-item (PHQ9) scale, min 0 max 27 with lower scores representing better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Jyoti Mishra, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- UC San Diego Health Psychiatry, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No